CLINICAL TRIAL: NCT06221449
Title: Effect of Lung Recruitment on Atelectasis in Lung-Healthy Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Lung Recruitment in Laparoscpic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Amany Said Abdel Haleem, Lecturer, Menoufia University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 7/2023ANET14
Record Dates: First submitted 2023-12-19; First posted 2024-01-24 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Atelectasis, Postoperative
Keywords: laparoscopic, atelectasis, recruitment maneuver,
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Intervention Model Description: comparison
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group (I) Control group:(31 patients) (Placebo Comparator): Patients will have controlled mechanical ventilation with these parameters (fixed Tidal Volume 6-8ml/Kg Ideal body weight - fixed fio2 0.5% - fixed POSITIVE end expiratory pressure 6 cm. water - fixed respiratory rate10-14 Respiratory rate /min)
  Interventions: Procedure: Positive end expiratory pressure
- Group (II) Sustained inflation group (SI): (31 patients) (Active Comparator): Patients will have controlled mechanical ventilation then after abdominal deflation, sustained inflation for 30 second by applying pressure 40 centimetreswater, with 5 these parameters (fixed Tidal Volume 6-8ml/Kg Ideal bogy weight - fixed fio2 0.5% - fixed positive end expiratory pressure 6 cmH2O - fixed respiratory rate 10-14 per minute.
  Interventions: Procedure: Positive end expiratory pressure
- Group (III) Stepwise PEEP increasing: (31 patients) (Active Comparator): Patients will have controlled mechanical ventilation, then after abdominal deflation gradual increasing in Positive end expiratory pressure 2 centimetres water every 5 respiratory cycle with maximum 10-12 centimetres water guided by hemodynamics & airway pressure not exceeding 40 centimetres water With these parameters (fixed Tidal Volume 6-8ml/Kg Ideal body weight - fixed fio2 0.5% -fixed respiratory rate10-14 .
  Interventions: Procedure: Positive end expiratory pressure

INTERVENTIONS:
Procedure: Positive end expiratory pressure — The patients will be divided into three groups:
  Control group:(31 patients); Patients will have controlled mechanical ventilation with these parameters (fixed Tidal Volume 6-8ml/Kg IBW - fixed fio2 0.5% - fixed PEEP 6 cmH2O - fixed respiratory rate10-14 RR/min) II) Group (II) Sustained inflation group (SI): (31 patients); Patients will have controlled mechanical ventilation then after abdominal deflation, sustained inflation for 30 second by applying pressure 40 cmH2O, with 5 these parameters (fixed Tidal Volume 6-8ml/Kg IBW - fixed fio2 0.5% - fixed PEEP 6 cmH2O - fixed respiratory rate 10-14 RR/min) III) Group (III) Stepwise PEEP increasing: (31 patients); Patients will have controlled mechanical ventilation, then after abdominal deflation gradual increasing in PEEP 2 cmH2O every 5 respiratory cycle with maximum 10-12 cmH2O guided by hemodynamics & airway pressure not exceeding 40 cmH2O.

SUMMARY:
The goal of this clinical trial study is to assess the effectiveness of different methods of lung recruitment maneuver on the incidence of atelectasis in adults undergoing laparoscopic cholecystectomy surgery using lung ultrasound Participants will be divided into three groups as: Control group, sustained inflation group (SI) and Stepwise Positive end expiratory pressure increasing group(Third group). Each contains 31 patients.

Control Group = Keep parameters all through the procedure without any changing GROUP(SI) = After abdominal deflation, we will apply sustained inflation by adjusting Adjustible pressure Limiting valve 40 centimetres water on spontaneous mode, holding the bag for 30 second.

Third group = After abdominal deflation, we will apply stepwise Positive Pressure increasing by 2 centimetres water every 5 breathing cycles till reaching 12 centimetres water and keeping it till extubation, with a maximum airway pressure not exceeding 40 centimetres water.

DETAILED DESCRIPTION:
the effectiveness of different methods of lung recruitment maneuver on the incidence of atelectasis in adults undergoing laparoscopic cholecystectomy surgery using lung ultrasound Participants will be divided into three groups as: Control group, sustained inflation group (SI) and Stepwise POSITIVE pressure increasing group. Each contains 31 patients.

Control Group = Keep parameters all through the procedure without any changing GROUP(SI) = After abdominal deflation, The investigators will apply sustained inflation by adjusting Adjustible pressure valve 40 centimetres water spontaneous mode, holding the bag for 30 second.

Third group = After abdominal deflation, the investigators will apply stepwise POSITIVE pressure increasing by 2 centimeters water 5 breathing cycles till reaching 12 centimetres water and keeping it till extubation, with a maximum airway pressure not exceeding 40 centimetreswater.

During the entire procedure the transducer head will be placed over one point of the chest selected by the operator where the area of atelectasis was detected The probe will be placed in the atelectasis area.

ELIGIBILITY:
Inclusion Criteria:

* Patients with healthy lungs

  * Age between 18 and 65 years old
  * Body mass index (BMI) <30 kg / m2
  * Physical status I-II of the American Society of Anesthesiologists (ASA)
  * Elective laparoscopic cholecystectomy.

Exclusion Criteria:

* Patient refusal
* Patients with preoperative ultrasound evidence of pulmonary atelectasis.
* Patients who will have conversion from laparoscopic to open surgery.
* Patients experiencing critical postoperative complications such as severe subcutaneous emphysema and pneumothorax.
* Patients with pulmonary, cardiac, and neuromuscular diseases and a corresponding surgical history and respiratory tract infections.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Incidence of atelectasis | one hour
  incidence

SECONDARY OUTCOMES:
Lung ultrasound score | one day
  0 no atelectasis with A lines
  1. multiple B lines
  2. white lung
  3. Lung consolidation
Blood pressure ( millimetre Mercury) | Two hour
  Measurements
Heart rate | Two hour
  Beat per minute
Hospital length of stay | One day
  Duration of stay at hospital in hours

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University, Shibīn al Kawm, Egypt